CLINICAL TRIAL: NCT07105319
Title: A Feasibility Study of Ropeginterferon for Treatment Free Remission in CML Patients Who Have a Sustained Deep Molecular Response
Brief Title: Ropeginterferon for Treatment Free Remission
Acronym: ROPEG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-Wook Kim (Other)
Responsible Party: Sponsor-Investigator, Dong-Wook Kim, Professor, Eulji University Hospital
Organization: Eulji University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UEMC-2021-09-025
Record Dates: First submitted 2025-04-18; First posted 2025-08-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: CML (Chronic Myelogenous Leukemia)
Keywords: Ropeginterferon; TFR; deep molecular response
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Intervention Model Description: This is a pilot randomized two-arm prospective study with/without Ropeginterferon in CML patients who have sustained MR4.5 for 24 months or more with TKIs The patients will be randomized to a ratio of 1:1 for each group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- randomized two-arm prospective study with/without Ropeginterferon in CML patients (Experimental): The patients will be randomized to a ratio of 1:1 for each group
  1. Investigational arm with Ropeginterferon (50 patients): Patients will be treated with 250 μg at week 0, 350 μg at week 2, and then 500 μg at week 4, and thereafter bi-weekly subcutaneous injection until week 24
  2. Comparator arm (50 patients): Patients will be followed with no further CML treatment
  Interventions: Drug: Ropeginterferon

INTERVENTIONS:
Drug: Ropeginterferon — 1. Investigational arm with Ropeginterferon (50 patients): Patients will be treated with 250 μg at week 0, 350 μg at week 2, and then 500 μg at week 4, and thereafter bi-weekly subcutaneous injection until week 24
  2. Comparator arm (50 patients): Patients will be followed with no further CML treatment

SUMMARY:
Ropeginterferon is a long-acting next-generation mono-pegylated interferon alfa-2b consisting of one isoform produced by PharmaEssentia Co. and the pegylated (PEG) formulations that require less frequent administration and have improved efficacy and tolerability.

In this study, patients in the investigational arm will receive Ropeginterferon subcutaneously with 250 μg at week 0, 350 μg at week 2, 500 μg at week 4, and thereafter 500 μg bi-weekly until week 24.

DETAILED DESCRIPTION:
This is a pilot, randomized, two-arm, prospective study with or without Ropeginterferon in CML patients who have sustained MR4.5 for 24 months or more with TKIs.

The patients will be randomized to either

1. Investigational arm with Ropeginterferon (50 patients): Patients will be treated with 250 μg at week 0, 350 μg at week 2, and then 500μg at week 4, and thereafter bi-weekly subcutaneous injection until week 24
2. Comparator arm (50 patients): Patients will be followed with no further CML treatment.

ELIGIBILITY:
Inclusion Criteria:

A patient must satisfy all the following criteria to be enrolled in the study.

1. New CML-CP at diagnosis
2. Patients aged 19 or more and 75 or less
3. BCR-ABL1 transcripts with e13a2 or e14a2 transcripts
4. Sustained MR4.5 for 24 months or more
5. Signed written informed consent

Exclusion Criteria:

* 1) Any contraindication to any of the interferon 2) Documented autoimmune disease at screening or in the medical history 3) Clinically relevant pulmonary infiltrates, pneumonia, and pneumonitis at screening 4) Systemic infections, e.g. hepatitis B, hepatitis C, or HIV at screening 5) Any investigational drug less than 6 weeks before the first dose of study drug or not recovered from effects of prior administration of any investigational agent 6) History or presence of depression requiring treatment with antidepressant 7) Any risk of suicide at screening or previous suicide attempts 8) Any significant morbidity or abnormality which may interfere with the study participation 9) Pregnancy and breast-feeding females of reproductive potential and males not using effective means of contraception 10) History of active substance or alcohol abuse within the last year 11) Evidence of severe retinopathy (e.g. cytomegalovirus retinitis, macular degeneration) or clinically relevant ophthalmological disorder (due to diabetes mellitus or hypertension) 12) Thyroid dysfunction not adequately controlled 13) History of major organ transplantation 14) History of uncontrolled severe seizure disorder 15) Leukocytopenia at the time of screening (count: < 4.0 x 109/L) 16) Thrombocytopenia at the time of screening (count: < 100 x 109/L) 17) History of other malignant diseases except for CML, including solid tumors and hematological malignancies (except basal cell and squamous cell carcinomas of the skin and carcinoma in situ of the cervix that has been completely excised and is considered cured) within the last 3 years

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Treatment-Free Remission (TFR) rates by 12 months after TKI discontinuation | the screening and week 4/8/12/16/20/24/32/40/48/60/ 72 then after every 12 weeks.
  To assess the preventive efficacy of Ropeginterferon in Major Molecular Response (MMR) loss after TKI discontinuation

CONTACTS AND LOCATIONS:
Locations (1):
- Eulji University Hospital, Uijeongbu-si, Gyeonggi-do, South Korea